CLINICAL TRIAL: NCT06847022
Title: Efficacy of Ultrasound-guided Transversalis Fascia Plane Block (TFPB) in Controlling Postoperative Pain After Transverse Incision in Gynecologic Surgery
Brief Title: Efficacy of US-guided Transversalis Fascia Plane Block (TFPB) in Controlling Postoperative Pain After Open Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, PREEYAPHAN ARUNAKUL, Assistant Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-AN-1-062/67
Record Dates: First submitted 2025-02-16; First posted 2025-02-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Transversalis Fascia Plane Block; Gynecologic Surgical Procedures
Keywords: Transversalis fascia plane block; open gynecologic surgery; transverse incision

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Patients in control group will receive general anesthesia for open gynecologic surgery.
- TFPB (Experimental): Patients in this study group will receive general anesthesia and US-guided bilateral TFPB after wound closure.
  Interventions: Procedure: US-guided transversalis fascia plane block

INTERVENTIONS:
Procedure: US-guided transversalis fascia plane block — US-guided bilateral transversalis fascia plane block, using Sonotap 110 mm and 0.25% bupivacaine 20 ml on each side, will be done after wound closure.
  Arms: TFPB

SUMMARY:
Transversalis fascia plane block (TFPB) has been studied and has shown to be very effective in controlling postoperative pain after caesarean section but has not been studied in open gynecologic surgery with transverse incision. Inadequate pain control after open gynecologic surgery is associated with negative consequences such as chronic pelvic pain. The investigators aimed to evaluate the efficacy of TFPB in controlling postoperative pain after open gynecologic surgery with transverse incision.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoing open gynecologic surgery under general anesthesia
* Age 18 - 70 years
* ASA Physical status I-III
* Transverse incision

Exclusion Criteria:

* Creatinine clearance is less than 30 ml/min
* Body weight < 50 kg
* Re-open surgery
* Persistent chronic pelvic pain
* Allergic to medications used in this study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study aims to evaluate pain after open gynecologic surgery, so only female are eligible.
Enrollment: 32 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Postoperative 24 hours morphine requirement | 24 hours

SECONDARY OUTCOMES:
postoperative pain score | 1 hour, 6 hours, 24 hours
Side effects from postoperative opioids | 24 hours
  nausea vomiting, itching, respiratory depression
Incidence of chronic pelvic pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Assist. Prof. Dr. Preeyaphan Arunakul, M.D., FRCAT, Principal Investigator — Faculty of Medicine, Thammasat University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Thammasat University, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Management of Chronic Pelvic Pain. In: Hibner M, editor. Management of Chronic Pelvic Pain: A Practical Manual. Cambridge: Cambridge University Press; 2021. p. i-ii.
- [Background] van Rijckevorsel DC, de Vries M, Schreuder LT, Wilder-Smith OH, van Goor H. Risk factors for chronic postsurgical abdominal and pelvic pain. Pain Manag. 2015;5(2):107-16. doi: 10.2217/pmt.14.47. PMID 25806905
- [Background] Chilkoti GT, Gaur D, Saxena AK, Gupta A, Agarwal R, Jain S. Ultrasound-guided transversalis fascia plane block versus wound infiltration for both acute and chronic post-caesarean pain management - A randomised controlled trial. Indian J Anaesth. 2022 Jul;66(7):517-522. doi: 10.4103/ija.ija_173_22. Epub 2022 Jul 22. PMID 36111099
- [Background] Black ND, Malhas L, Jin R, Bhatia A, Chan VWS, Chin KJ. The analgesic efficacy of the transversalis fascia plane block in iliac crest bone graft harvesting: a randomized controlled trial. Korean J Anesthesiol. 2019 Aug;72(4):336-343. doi: 10.4097/kja.d.18.00352. Epub 2019 Mar 19. PMID 30886131
- [Background] Fouad AZ, Abdel-Aal IRM, Gadelrab MRMA, Mohammed HMES. Ultrasound-guided transversalis fascia plane block versus transmuscular quadratus lumborum block for post-operative analgesia in inguinal hernia repair. Korean J Pain. 2021 Apr 1;34(2):201-209. doi: 10.3344/kjp.2021.34.2.201. PMID 33785672
- [Background] Geng ZY, Zhang Y, Bi H, Zhang D, Li Z, Jiang L, Song LL, Li XY. Addition of preoperative transversus abdominis plane block to multimodal analgesia in open gynecological surgery: a randomized controlled trial. BMC Anesthesiol. 2023 Jan 12;23(1):21. doi: 10.1186/s12871-023-01981-w. PMID 36635627
- [Background] Wilson SH, Hellman KM, James D, Adler AC, Chandrakantan A. Mechanisms, diagnosis, prevention and management of perioperative opioid-induced hyperalgesia. Pain Manag. 2021 Apr;11(4):405-417. doi: 10.2217/pmt-2020-0105. Epub 2021 Mar 29. PMID 33779215
- [Background] VanDenKerkhof EG, Hopman WM, Goldstein DH, Wilson RA, Towheed TE, Lam M, Harrison MB, Reitsma ML, Johnston SL, Medd JD, Gilron I. Impact of perioperative pain intensity, pain qualities, and opioid use on chronic pain after surgery: a prospective cohort study. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):19-27. doi: 10.1097/AAP.0b013e318237516e. PMID 22157741
- [Background] Ohnesorge H, Gunther V, Grunewald M, Maass N, Alkatout I. Postoperative pain management in obstetrics and gynecology. J Turk Ger Gynecol Assoc. 2020 Dec 4;21(4):287-297. doi: 10.4274/jtgga.galenos.2020.2020.0024. Epub 2020 Jun 5. PMID 32500680
- [Background] Amberbir WD, Bayable SD, Fetene MB. The prevalence and factors associated with acute postoperative pain in elective gynecologic surgical patients at two referral hospitals in Addis Abeba, Ethiopia, 2021: a cross-sectional study. Ann Med Surg (Lond). 2023 Apr 27;85(6):2506-2511. doi: 10.1097/MS9.0000000000000716. eCollection 2023 Jun. PMID 37363541
- [Background] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Background] Pinarbasi A, Altiparmak B, Korkmaz Toker M, Pirincci F, Ugur B. Ultrasound-guided transversalis fascia plane block or transversus abdominis plane block for recovery after caesarean section: A randomised clinical trial. Eur J Anaesthesiol. 2024 Oct 1;41(10):769-778. doi: 10.1097/EJA.0000000000002041. Epub 2024 Jul 22. PMID 39039833